CLINICAL TRIAL: NCT00480857
Title: Salvage Radiation Therapy and Docetaxel (Taxotere) for Biochemical Failure After Radical Prostatectomy
Brief Title: Salvage Radiation Therapy and Taxotere for PSA Failure After Radical Prostatectomy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding.
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2006.066; HUM 7093 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2007-05-29; First posted 2007-05-31 (Estimated); Results first posted 2015-01-16 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-09

CONDITIONS: Prostate Cancer
Keywords: Prostate; Radiation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel (Experimental)
  Interventions: Drug: Docetaxel (Taxotere)

INTERVENTIONS:
Drug: Docetaxel (Taxotere) — Concurrent weekly docetaxel at 20mg/m2 with radiation therapy. Chemo dose may be held or reduced based on specific lab parameters.

SUMMARY:
The main purpose of this study is to try to find out whether adding chemotherapy to the standard treatment for your stage of prostate cancer is more effective than the standard treatment by itself. The kind of treatment that most physicians would consider standard for this stage of prostate cancer is radiation therapy alone, possibly in combination with hormonal therapy. In this study, all patients will receive chemotherapy and radiation therapy. It is hoped that chemotherapy will be found to provide additional benefit, but chemotherapy has significant side effects. The use of chemotherapy is experimental in prostate cancer; it needs to be tested to determine if it is beneficial and to find out more about the side effects of the two different treatments. This study is to determine the effects, good and/or bad, of adding chemotherapy to radiation therapy as "salvage" treatment for recurrent prostate cancer after surgery.

DETAILED DESCRIPTION:
There is no treatment proven more effective for clinically localized prostate cancer than radical prostatectomy. Nonetheless, approximately 30,000 men annually in the U.S. develop recurrence of their prostate cancer after prostatectomy. Radiation therapy is commonly utilized as attempted salvage treatment for patients who develop a rising PSA (Prostate Specific Antigen) after prostatectomy and have no evidence of metastatic disease. This study is designed to determine whether concurrent chemotherapy, weekly docetaxel, and daily radiation therapy will result in improved disease control and survival rates over those obtained with radiotherapy alone in the treatment of men with biochemical recurrence after radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Performance Status: Karnofsky performance status ≥ 80% (Performance status is an attempt to quantify cancer patients' general well-being and activities of daily life. The Karnofsky score runs from 100 to 0, where 100 is "perfect" health and 0 is death.)
* Has undergone prostatectomy for histologically confirmed adenocarcinoma of the prostate at least 6 weeks prior to registration. (If prostatectomy was completed at an outside facility, a University of Michigan pathology review must take place to confirm adenocarcinoma.)
* Has biochemical evidence of failure as determined by at least two PSA measurements after prostatectomy. This must be demonstrated by an increase of at least 0.1 ng/mL between two consecutive measurements, both obtained after prostatectomy. The most recent measurement (within 28 days of registration) must be 0.3 ng/mL or greater.
* Has undergone pelvic CT (Computerized Tomography) scan and radionuclide bone scan within 90 days prior to registration that showed no evidence of regional or distant nodal or bone metastasis.
* Patients with pelvic or abdominal lymph nodes equivocal or questionable by imaging are eligible if the nodes are < 1.5 cm in long axis.
* Equivocal bone scan findings are allowed if plain films show no conclusive evidence of metastasis.
* Hematologic Criteria: CBC (Complete Blood Count)/differential obtained within 28 days prior to registration on study, with adequate bone marrow function defined as follows:

  * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
  * Platelets ≥ 100,000 cells/mm3
  * Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb = 8.0 g/dl is acceptable).
* Hepatic Criteria within 28 days prior to registration:

  * Total bilirubin < 1 x institutional upper limit of normal (ULN)
  * ALT (Alanine Transaminase), AST (Aspartate Aminotransferase), and alkaline phosphatase must be within the eligible ranges stipulated in protocol table
  * Serum creatinine < 2 x ULN
* Both radiation oncology and medical oncology consultation prior to registration.
* Pharmacologic androgen ablation for prostate cancer will be allowed only if given prior to prostatectomy.
* Patient must sign study specific informed consent prior to study entry.
* Peripheral neuropathy: must be ≤ grade 1
* Patients must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.

Exclusion Criteria:

* Patients with a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80.
* Evidence of M1 metastatic disease
* Pathologically positive lymph nodes or nodes > 1.5 cm on imaging
* Prior pelvic radiotherapy that would result in overlap of radiation therapy fields or systemic cytotoxic chemotherapy.
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 5 years (for example,carcinoma in situ of the oral cavity or bladder are permissible)
* Severe, active co-morbidity, defined as follows, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the 6 months prior to registration.
  * Transmural myocardial infarction within the 6 months prior to registration
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-03; Primary Completion 2013-08 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A. Hamstra, M.D., Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Jackson WC, Feng FY, Daignault S, Hussain M, Smith D, Cooney K, Pienta K, Jolly S, Hollenbeck B, Olson KB, Sandler HM, Ray ME, Hamstra DA. A phase 2 trial of salvage radiation and concurrent weekly docetaxel after a rising prostate-specific antigen level after radical prostatectomy. Adv Radiat Oncol. 2015 Dec 9;1(1):59-66. doi: 10.1016/j.adro.2015.11.001. eCollection 2016 Jan-Mar. PMID 28799570

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Docetaxel
Started | 19
Completed | 17
Not Completed | 2
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Docetaxel
Number analyzed (Participants) | 19
Age, Continuous [Mean (Full Range); unit: years] | 66 [43 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Alive Without Progression at 4 Years
Description: The primary objective is to assess the 4-year progression free proportion of patients treated with concurrent weekly docetaxel (TAXOTERE) and salvage prostate bed radiation therapy among patients with biochemical recurrence after radical prostatectomy.
Time Frame: 4 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Docetaxel
Number analyzed (Participants) | 19
percentage of patients | 42 [24 to 60]

2. Secondary Outcome: Number of Patients That Achieve a Post-radiotherapy PSA Nadir of 0.1 ng/mL or Less
Description: To determine the rates of complete biochemical response (as defined by achievement of a post-radiotherapy PSA nadir of 0.1 ng/mL or less) after concurrent weekly docetaxel (TAXOTERE) and salvage prostate bed radiation therapy.
Time Frame: 4 years
Measure: Number; unit: patients
Arm/Group | Docetaxel
Number analyzed (Participants) | 19
patients | 12

3. Secondary Outcome: The Percentage of Patients That Experience at Least 1 Grade 1, 2, 3 and 4 Toxicities
Description: To determine the rates of toxicities among patients treated with concurrent weekly docetaxel (TAXOTERE) and salvage prostate bed radiation therapy.
  G1 events are considered mild. G2 events are considered moderate G3 events are considered severe G4 events are considered life-threatening
Time Frame: 4 years
Measure: Number; unit: percentage of patients
Arm/Group | Docetaxel
Number analyzed (Participants) | 19
percentage of patients
  Patients that experience at least 1 G1 toxicity | 79
  Patients that experience at least 1 G2 toxicity | 50
  Patients that experience at least 1 G3 toxicity | 58
  Patients that experience at least 1 G4 toxicity | 11

4. Secondary Outcome: The Number of Patients That Experience Evidence of Local Recurrence
Description: The number of patients that have local disease recurrence by imaging and clinical findings.
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel
Number analyzed (Participants) | 19
Participants | 0

5. Secondary Outcome: The Number of Patients Alive
Description: The number of patients alive at 4 years.
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel
Number analyzed (Participants) | 19
Participants | 18

ADVERSE EVENTS:
Arm/Group | Docetaxel
Serious Adverse Events (participants affected / at risk) | 6/19
Other Adverse Events (participants affected / at risk) | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel (N=19)
Lymphopenia (Blood and lymphatic system disorders) | 4
Upper Gastrointestinal Bleed (Gastrointestinal disorders) | 1
Hematochezia (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel (N=19)
Fatigue (General disorders) | 14
Bowel Frequency/Urgency (Gastrointestinal disorders) | 8
Urinary Frequency/Urgency (Renal and urinary disorders) | 6
Other (General disorders) | 3
Hematochezia (Gastrointestinal disorders) | 3
Neuropathy (Nervous system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Anemia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 14
Rectal (Gastrointestinal disorders) | 4
Weights Loss (General disorders) | 1
Upper GI Bleed (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes